CLINICAL TRIAL: NCT05715788
Title: Prone Positioning Versus Prone Positioning and NO Inhalation in COVID-19 Associated Acute Respiratory Distress Syndrome.
Brief Title: Prone Positioning vs. Prone Positioning and NO Inhalation in COVID-19 ARDS.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ppv-vs-ppvno
Record Dates: First submitted 2023-02-04; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Nitric Oxide; Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients ventilated in prone position: Patients ventilated in prone position
  Interventions: Behavioral: prone positioning
- Patients ventilated in prone position with NO inhalation: Patients ventilated in prone position with NO inhalation
  Interventions: Drug: Nitric oxide; Behavioral: prone positioning

INTERVENTIONS:
Drug: Nitric oxide — Nitric oxide inhalation at 20 ppm
  Groups: Patients ventilated in prone position with NO inhalation
Behavioral: prone positioning — vatilation in prone position
  Other Names: PPV

SUMMARY:
The investigators aim to investigate the effects of prone positioning and prone positioning with NO inhalation for COVID-19 patients with ARDS.

DETAILED DESCRIPTION:
The investigators aim to investigate the effects of prone positioning and prone positioning with NO inhalation for COVID-19 patients with ARDS. Patients with COVID-19-associated ARDS were ventilated in prone position with or without NO inhalation, the arterial blood gas (ABG) tests were performed at 16 hours after prone positioning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with COVID-19 associated ARDS

Exclusion Criteria:

* patients who have contraindication for prone positioning, including pregnant, post-abdomen surgery within a week; hypercapnic respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 associated ARDS
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
P/F ratio | 16 hours
  P/F ratios in each group

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No